CLINICAL TRIAL: NCT02683681
Title: Heart Failure Intraoperative Tissue Sample Acquisition Registry
Brief Title: HF Tissue Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Drakos Lab, University of Utah Eccles Institute for Human Genetics (Unknown); Center for Molecular and Genetic Research, LDS Hospital Cardiovascular Genetics Lab (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1009557
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — * Tissue samples will be obtained at the time of LVAD implantation by keeping the part of the left ventricular apex that the surgeon is removing in order to place the inflow cannula of the LVAD. No extra tissue sample other than the tissue that has to be removed as a part of a standard LVAD operation needs to be obtained.
  * Tissue samples will be acquired from the failing heart at the time of heart transplantation, after it has been excised and a donor heart has been implanted in its place.
  * Control tissue samples will be acquired intraoperatively during cardiac surgery wherein any amount of excised tissue is routinely discarded.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry study. This is an observational, non-randomized, open, long-term project to collect biological samples (e.g. tissue and blood samples) in addition to clinical information and laboratory test results, from end-stage patients who undergo LVAD implantation and/or heart transplantation. There are no investigational treatments, drug or procedures associated with participation in registry activities.

Data collection will not immediately influence the course of treatment for any patient.

DETAILED DESCRIPTION:
After informed consent is obtained from the patient, the blood samples will be obtained either during a procedure from access lines inserted for the procedure or they will be drawn when other ordered lab work is done at specific time points. While blood samples collection is preferred, it is not required, and the decision to collect blood samples will be left to the discretion of the investigator.

* Tissue samples will be obtained at the time of LVAD implantation by keeping the part of the left ventricular apex that the surgeon is removing in order to place the inflow cannula of the LVAD. No extra tissue sample other than the tissue that has to be removed as a part of a standard LVAD operation needs to be obtained.
* Tissue samples will be acquired from the failing heart at the time of heart transplantation, after it has been excised and a donor heart has been implanted in its place.
* Control tissue samples will be acquired intraoperatively during cardiac surgery wherein any amount of excised tissue is routinely discarded.

In some cases, when a patient has an existing LVAD implant for destination therapy, and is not eligible for cardiac transplant, and is not scheduled for cardiac surgery in the foreseeable future, the patient will be approached for consent for blood samples. In addition, consent to obtain intraoperative tissue samples is requested in the event cardiac surgery occurs and/or the device is explanted for any reason in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be in one of the following groups:

   1.1. Patients must be eligible for a -
   * LVAD implantation or
   * Heart transplantation 1.2. Patients must be scheduled for another type of cardiac surgery during which tissue is excised that would normally be discarded after surgery.

   1.3. Patients must have a VAD already implanted as destination therapy with no cardiac surgery scheduled at the time of consent.
2. Patients must agree to one or more blood and/or cardiac tissue sample donation(s), and longterm storage of these biological samples.
3. Patients must be > 18 years of age.

Exclusion Criteria:

Patients will be excluded from the study if any of the following conditions are present:

1. The patient or the patient's personal representative is unable or unwilling to give written informed consent for participation.
2. Patients who are less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seen at participating facilities for left ventricular assist device (LVAD) implantation and/or heart transplantation will be screened for this registry study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 20 years

IPD SHARING:
Plan to Share IPD: No